CLINICAL TRIAL: NCT04150562
Title: Phase II Trial of Avelumab (Bavencio) With IL-15 in Subjects With Clear-Cell Renal Carcinoma
Brief Title: Avelumab (Bavencio) With IL-15 in Subjects With Clear-Cell Renal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to manufacturer withdrawal of support (study medication) due to lack of enrollment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200007; 20-C-0007
Record Dates: First submitted 2019-11-01; First posted 2019-11-04 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Clear-Cell Renal Carcinoma
Keywords: Antibody Dependent Cellular Cytotoxicity (ADCC); Anti-PD-L1 monoclonal antibody
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Interleukin-15; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1- Experimental Treatment: Safety Run-in (Experimental): Interleukin 15 (IL-15) by continuous intravenous (CIV) infusion at escalating doses of 2 and 4 mcg/kg/day on days 1-5 of each 28-day cycle (max 4 cycles) with avelumab by intravenous (IV) infusion at a dose of 800mg on Day 8 and 22 of each cycle
  Interventions: Drug: rhIL-15; Biological: Avelumab
- Arm 2-Experimental Treatment: Dose Expansion (Experimental): Interleukin 15 (IL-15) by continuous intravenous (CIV) infusion at 4 mcg/kg/day on days 1-5 of each 28- day cycle (max 4 cycles) with avelumab by intravenous (IV) infusion at a dose of 800mg on Day 8 and 22 of each cycle
  Interventions: Drug: rhIL-15; Biological: Avelumab

INTERVENTIONS:
Drug: rhIL-15 — Recombinant human Interleukin-15 (rhIL-15) will be administered by continuous intravenous infusion (CIV) at a starting dose of 2 mcg/kg/day for the first dose level followed by a second dose level of 4mcg/kg/day on days 1-5 of the 28-day cycle of each of four cycles.
  Other Names: Recombinant human Interleukin-15
Biological: Avelumab — avelumab (800mg by intravenous (IV) will be administered on days 8 and 22 of the 28- day cycle for four cycles
  Other Names: Bavencio

SUMMARY:
Background:

-Clear-cell renal cell carcinoma (ccRCC) is a kind of kidney cancer. The drug avelumab may help direct the immune response to the tumors and can prolong the immune response. The drug Interleukin-15 (IL-15) stimulates certain kinds of white blood cells that have the potential to attack the cancer.

Objective:

-To test whether IL-15 and avelumab administered together are safe and effective at treating ccRCC.

Eligibility:

-People ages 18 and older with relapsed, metastatic biopsy proven clear cell renal cell carcinoma (ccRCC) that has not responded to standard treatments

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, heart, and lung tests
* Computed tomography (CT) and positron emission tomography (PET) scans and possible MRI: Participants will lie in a machine that takes pictures of the body. For the CT scan, they may receive an oral contrast agent by mouth and normally receive IV contrast through a vein to improve the x-ray images.
* Tumor sample to confirm expression of avelumab target: If one is not available, participants will require a new biopsy that is generally obtained by a needle that is inserted into the tumor.

Participants will get the study drugs by vein for up to four 28-day cycles. The IL-15 will be given through a vein continuously for the first 5 days (120 hours) of each cycle. They avelumab will be given through a vein over about 1 hour on days 8 and 22 of each cycle. Participants will be hospitalized for their 1st week of IL-15 cycle and may be able to receive their subsequent IL-15 treatment as an outpatient depending on their side effects. Participants who receive the infusion as an outpatient will return to the hospital each day for a new bag of IL-15. Participants who cannot or do not want to be treated as an outpatient will be treated in the hospital during their 5-day IL-15 infusions.

* Participants will need a midline venous catheter which is longer than a standard venous catheter but is still inserted into a peripheral vein in their arm.
* Participants will have repeats of blood tests to monitor the blood counts and chemistry throughout the study.
* Participants will have follow-up visits 30 days after their last treatment, every 60 days for the first 6 months, every 90 days for 2 years, then every 6 months.

DETAILED DESCRIPTION:
Background:

* Clear-cell renal cell carcinoma (ccRCC) is among the 10 most frequent diagnostic cancers in the United States with more than an estimated 62,000 new cases in 2016. The prognosis for patients with metastatic disease is poor with survival rates of 8%.
* The immunologic effects of recombinant human Interleukin-15 (rhIL-15), a stimulatory cytokine that promotes the differentiation and activation of NK cells, monocytes and long term cluster of differentiation 8 (CD8)+ memory T-cells, has been assessed in several Phase 1 trials in cancer patients.
* Avelumab is an anti-programmed death ligand-1 (PD-L1) fully human immunoglobulin G1 (IgG1) antibody that inhibits programmed cell death protein 1 (PD1)/PD-L1 interactions while leaving the PD1/Programmed cell death 1 ligand 2 (PD-L2) pathway intact and enhances immune activation against tumor cells. It has received United States (U.S.) Food and Drug Administration (FDA) accelerated approval for the treatment of patients with metastatic Merkel cell carcinoma (MCC) and urothelial carcinoma.
* Unlike other approved anti-PD-L1/PD1 antibodies, avelumab induces lysis of tumor cells via antibody-dependent cell-mediated cytotoxicity (ADCC), indicating an additional mechanism of action. However, avelumab has not shown ADCC against normal immune cell subsets in humans.
* More than 50% of ccRCC is PD-L1+ with higher expression in unfavorable prognostic tumors. Since the anti-PD-L1 antibody avelumab has shown ADCC activity in vitro, agents that may enhance ADCC by increasing number and activity of Fc-binding effector cells -such as recombinant human Interleukin-15 (rhIL-15) - could improve efficacy of avelumab in this disease.

Objectives:

-Determine the efficacy of combined continuous intravenous infusion (CIV) rhIL-15 and avelumab treatment in patients with anti-PD-1/PD-L1 refractory metastatic clear cell renal carcinoma (ccRCC) by assessing the overall response rate

Eligibility:

* Age greater than or equal to 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1
* Histologically proven metastatic clear cell renal carcinoma with greater than or equal to 5% expression of PD-L1 in the tumor area confirmed by immunohistochemistry (IHC)
* Patients must have failed or relapsed and have progressive disease after at least 2 prior therapies that include multityrosine kinase inhibitor like axitinib or sunitinib and an anti-PD1 or PD-L1 immune checkpoint inhibitor therapy like nivolumab which could have been administered in combination with an anti-cluster of differentiation 152 (CTLA4) agent like ipilimumab
* Adequate organ and marrow function

Design:

* Open-label, single-center, non-randomized Phase II study
* Safety Run-in Cohort with 3-6 patients at dose level 2mcg/kg and 4mcg/kg continuous intravenous (CIV) interleukin-15 (IL-15) (recommended phase II dose) will ensure safety of recommended phase II dose rhIL-15 with fixed dose avelumab with Dose Expansion Cohort at 4mcg/kg dose level
* Efficacy of the combination will be assessed in a Simon two-stage phase II design with 9 or 17 patients depending on demonstration of clinical activity in the initial group of 9 patients
* Maximum 4 cycles (28-day cycle) of combination therapy
* To explore both Safety Run-in Cohort and further evaluation in a Dose Expansion Cohort, the accrual ceiling will be set at 25 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically proven metastatic clear cell renal carcinoma with greater than or equal to 5% expression of programmed death-ligand 1 (PD-L1) on the tumor cells confirmed by immunohistochemistry (IHC) in the national Cancer Institute (NCI) Lab of Pathology. Archival tumor sample may be used but if archival tissue is not available or is not adequate, tissue biopsy will be required.
* Patients must have failed or relapsed and have progressive disease after at least 2 prior therapies that include multityrosine kinase inhibitor (mTKI) like axitinib or sunitinib and an anti-Programmed cell death protein 1 (PD1) or PD-L1 (ICI) therapy like nivolumab which could have been administered in combination with an anti-cluster of differentiation 152 (CTLA4) agent like ipilimumab. Patients who received an immune checkpoint inhibitor (ICI) in combination with a mTKI would be eligible for the trial if they received another appropriate treatment. Adjuvant or neoadjuvant with either type of agent would not fulfill this requirement only treatment for metastatic disease will be considered to satisfy this criterion.
* Disease must be measurable with at least one measurable lesion by the Response Evaluation Criteria in Solid Tumors (Recist) v1.1 criteria that is different from the lesion biopsied.
* Age >=18 years

NOTE: Because no dosing or adverse event data are currently available on the use of recombinant human Interleukin-15 (rhIL-15) in combination with avelumab in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials

* Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky >=80%)
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * absolute lymphocyte count greater than or equal to 500/mcL
  * Hemoglobin greater than or equal to 10 g/dL
  * Platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional ULN
  * Serum creatinine less than or equal to 1.5 X institutional ULN

OR

* Creatinine clearance greater than or equal to 50 mL/min/1.73 m^2 for patients with creatinine levels >1.5 institutional ULN
* Negative serum or urine pregnancy test at screening for women of childbearing potential (WOCBP).

NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. WOCBP must have a negative pregnancy test (human chorionic gonadotropin (HCG) blood or urine) during screening.

* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 1 month after completion of rhIL-15 and avelumab administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C).
* Persisting toxicity related to prior therapy of grade > 1, with the exception of the following: alopecia, sensory neuropathy grade <= 2, or other grade <= 2 not constituting a safety risk based on investigator's judgement.
* Patients who are receiving any other investigational agents
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses <= 10 mg/day of prednisone or equivalent; or,
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication).
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with previous malignant disease other than the target malignancy within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
* Patients with history of any organ transplantation
* Vaccination within 4 weeks of the first dose of avelumab. Vaccination with a live vaccine while on trial is prohibited.

NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to rhIL-15 or avelumab.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding. Based on its mechanism of action, avelumab can cause fetal harm when administered to a pregnant woman. Animal studies have demonstrated that inhibition of the PD-1/PD-L1 pathway can lead to increased risk of immune-mediated rejection of the developing fetus resulting in fetal death. These potential risks may also apply to other agents used in this study.
* Patients with active bacterial infections, documented human immunodeficiency virus (HIV) infection or positive screening serology, polymerase chain reaction (PCR) evidence for active or chronic hepatitis B or hepatitis C, or positive screening hepatitis B virus (HBV)/hepatitis C virus (HCV) serology without documentation of successful curative treatment
* Patients with active or history of any autoimmune disease, including asthma requiring chronic inhaled or oral corticosteroids, or with history of asthma requiring mechanical ventilation; patients with a history of mild asthma that are on or can be switched to non-corticosteroid bronchodilator regimens are eligible
* Cardiovascular disease: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Waldmann TA, Dubois S, Miljkovic MD, Conlon KC. IL-15 in the Combination Immunotherapy of Cancer. Front Immunol. 2020 May 19;11:868. doi: 10.3389/fimmu.2020.00868. eCollection 2020. PMID 32508818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0007.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Arm 1 Safety Run-In Dose Level 2 at 4 mcg/kg/day due to early study closure. No participants were enrolled on the Arm 2 Dose Expansion group.
Groups:
- Arm 1- Safety Run-in Dose Level 1: Interleukin 15 (IL-15) by continuous intravenous (CIV) infusion at 2 mcg/kg/day on days 1-5 of each 28-day cycle (max 4 cycles) with avelumab by intravenous (IV) infusion at a dose of 800mg on Day 8 and 22 of each cycle
- Arm 2-Dose Expansion: Interleukin 15 (IL-15) by continuous intravenous (CIV) infusion at 4 mcg/kg/day on days 1-5 of each 28- day cycle (max 4 cycles) with avelumab by intravenous (IV) infusion at a dose of 800mg on Day 8 and 22 of each cycle to determine efficacy of treatment.
Period: Overall Study
Arm/Group | Arm 1- Safety Run-in Dose Level 1 | Arm 2-Dose Expansion
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.75 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete Response + Partial Response)
Description: Response was assessed using the Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST)v1.1. Immune related complete response (irCR) is at least two radiographic determinations of complete response (CR - e.g., disappearance of all target lesions) at least 4 weeks apart and before Immune related progressive disease (irPD - defined as at least two consecutive radiographic determinations of progressive disease ((PD - e.g., appearance of one or more new lesions) at least 4 weeks apart). at least 4 weeks apart). Immune related partial response (irPR) is at least two radiographic determinations of partial response (PR - e.g., 30% decrease of target lesions) or better at least 4 weeks apart and before irPD (and not qualifying for an irCR).
Time Frame: Following start of study medication while on treatment, approximately 2 months.
Measure: Number; unit: proportion of participants
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
proportion of participants
  Immune related complete response (irCR) | 0
  Immune related partial response (irPR) | 0

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from the initial response (irCR, irPR or irSD) to progression or death, whichever comes first. Response was assessed using the Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST)v1.1. Immune related complete response (irCR) is at least two radiographic determinations of complete response (CR) at least 4 weeks apart and before Immune related progressive disease (irPD - defined as at least two consecutive radiographic determinations of progressive disease (PD) at least 4 weeks apart). Immune related partial response (irPR) is at least two radiographic determinations of partial response (PR) or better at least 4 weeks apart and before irPD (and not qualifying for an irCR). Immune related stable disease (irSD) is at least one radiographic assessment of stable disease (SD) (or better) ≥ 6 weeks after the first trial treatment administration and before irPD (and not qualifying for irCR or irPR).
Time Frame: Following start of study medication while on treatment, up to 1-2 months.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
Days | 13 [0 to 26]

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever comes first. Progression was assessed using the Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST)v1.1. Immune related progressive disease (irPD) is defined as at least two consecutive radiographic determinations of progressive disease (PD - e.g., appearance of one or more new lesions) at least 4 weeks apart).
Time Frame: Monitoring frequency is every two cycles through completion of study then annually until progressive disease is noted, an average of 73 days.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
Days | 73 [62 to 84]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of study enrollment until time of death from any cause.
Time Frame: time from the date of study enrollment until time of death from any cause, an average of 167 days
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
Days | 167 [147 to 187]

5. Secondary Outcome: Number of Grade 3 Adverse Events Possibly, Probably or Definitely Related to Treatment of rhIL-15 + Avelumab
Description: Adverse events were assessed using the Common Terminology Criteria for Adverse Events (CTCAE)v5.0. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse events.
Time Frame: 4 cycles (each cycle is 28 days), up to 112 days
Measure: Number; unit: adverse events
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
adverse events
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 13 months and 24 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1- Safety Run-in Dose Level 1
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 13 months and 24 days.
Arm/Group | Arm 1- Safety Run-in Dose Level 1
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Safety Run-in Dose Level 1 (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- Safety Run-in Dose Level 1 (N=2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (2)
Flu like symptoms (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (6)
Nausea (Gastrointestinal disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT04150562/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT04150562/ICF_001.pdf